CLINICAL TRIAL: NCT00539188
Title: A Double-Blind, Placebo-controlled Pilot Study of NAC Addition to Dialectical Behavioral Therapy for the Treatment of Self-Injurious Behavior Associated With Borderline Personality Disorder
Brief Title: N-Acetylcysteine in Adjunct to DBT for the Treatment of Self-Injurious Behavior in BPD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to poor subject compliance.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0610001908
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Borderline Personality Disorder; Self-Injurious Behavior
Keywords: Borderline Personality Disorder(BPD); Dialectical Behavioral Therapy (DBT); glutamate; N-Acetylcysteine; Borderline Personality Disorder with Self-Injurious Behavior
MeSH Terms: conditions — Borderline Personality Disorder; Self-Injurious Behavior | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): Patients randomized to this arm will receive N-Acetylcysteine augmentation, at a standard dose (3000 mg daily), in addition to the medication regimen they are on at enrollment
  Interventions: Drug: N-Acetylcysteine
- placebo (Placebo Comparator): Patients randomized to this arm will receive placebo, formulated to be indistinguishable from N-Acetylcysteine, in addition to the medication regimen they are on at study enrollment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 3000 mg PO (1200 mg AM, 1800 mg PM), 6 weeks
  Other Names: NAC
  Arms: N-Acetylcysteine
Drug: placebo — placebo, 2 capsules PO AM, 3 capsules PO PM, 6 weeks
  Arms: placebo

SUMMARY:
Self-Injurious Behavior (SIB) is a dangerous and common symptom in Borderline Personality Disorder (BPD) patients. Approximately 70% of patients with BPD engage in SIB at some point, compared to 17.5% of patients with other personality disorders. While SIB may prompt unnecessary psychiatric hospitalizations, it may also cause potential underestimation of the lethality of suicidal behavior, thus creating a major and confusing challenge in the practice of clinical psychiatry.

Dialectical Behavioral Therapy (DBT) is a collection of therapeutic techniques focused on emotional regulation, impulse control, and improving safety in patients with BPD and others with marked self-destructive behavioral tendencies. Though DBT has marked ability to reduce BPD symptomatology, including SIB, improvement in SIB is limited and dependent on extensive therapy and time.

Furthermore, the literature on the pharmacological treatment of SIB associated with BPD is scarce. Animal studies suggest that SIB may be associated with an imbalance between dopamine and glutamate in the brain. Anti-seizure medications that modulate glutamate transmission, such as lamotrigine and topiramate, have been suggested to be effective in the treatment of SIB in humans.

Preliminary evidence suggests that antiglutamatergic medications may decrease SIB in patients with BPD. Early studies have focused on the antiglutamatergic drug riluzole. More recently, we have become interested in the amino acid N-acetylcysteine (NAC), which is used clinically for its antioxidant properties and is widely available as a nutritional supplement. Recent animal studies have suggested that NAC can modulate glutamate in the central nervous system in a way very similar to that proposed for riluzole, and indeed we have observed NAC to have an effect similar to riluzole in a case of treatment-refractory obsessive-compulsive disorder.

This study will be a double-blind, randomized, and placebo-controlled evaluation of N-Acetylcysteine as an adjunct to DBT in the treatment of SIB associated with BPD. Subjects participating in this study will be recruited exclusively from the Dialectical Behavioral Therapy program of the Yale-New Haven Hospital, in order to maximize homogeneity of the psychotherapeutic care received during their participation.

DETAILED DESCRIPTION:
Investigators have withdrawn study due to poor subject compliance. After 3 consecutive participants were either unable to complete all 6 weeks of the study or dropped out of the DBT program, a decision was reached to discontinue recruitment and study was terminated.

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder, as assessed by SCID-II
* A score of 10 or greater on the Self Harm Inventory (SHI) at time of evaluation
* Ability to give informed consent
* agreement to engage in a reliable form of birth control (women only)

Exclusion Criteria:

* primary diagnosis of a psychotic disorder
* active substance abuse or dependence
* unstable medical condition
* History of intolerance/allergic reaction to N-Acetylcysteine
* pregnancy, breastfeeding, or intent to become pregnant during study
* Inability to understand English
* Cognitive Impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Pittenger, MD,PhD, Principal Investigator — Yale University
Locations (1):
- Yale OCD Research Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Background] Coric V, Taskiran S, Pittenger C, Wasylink S, Mathalon DH, Valentine G, Saksa J, Wu YT, Gueorguieva R, Sanacora G, Malison RT, Krystal JH. Riluzole augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. Biol Psychiatry. 2005 Sep 1;58(5):424-8. doi: 10.1016/j.biopsych.2005.04.043. PMID 15993857
- [Background] Pittenger C, Krystal JH, Coric V. Glutamate-modulating drugs as novel pharmacotherapeutic agents in the treatment of obsessive-compulsive disorder. NeuroRx. 2006 Jan;3(1):69-81. doi: 10.1016/j.nurx.2005.12.006. PMID 16490414
- [Background] Smith BD. Self-mutilation and pharmacotherapy. Psychiatry (Edgmont). 2005 Oct;2(10):28-37. PMID 21120088
- [Background] Linehan MM (1993). The Cognitive-Behavioral Treatment of Borderline Personality Disorder. New York: The Guilford Press.
- [Background] Pittenger C, Bloch MH, Williams K. Glutamate abnormalities in obsessive compulsive disorder: neurobiology, pathophysiology, and treatment. Pharmacol Ther. 2011 Dec;132(3):314-32. doi: 10.1016/j.pharmthera.2011.09.006. Epub 2011 Sep 22. PMID 21963369

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine: Patients randomized to this arm will receive N-Acetylcysteine augmentation, at a standard dose (3000 mg daily), in addition to the medication regimen they are on at enrollment
  N-Acetylcysteine : 3000 mg PO (1200 mg AM, 1800 mg PM), 6 weeks
- Placebo: Patients randomized to this arm will receive placebo, formulated to be indistinguishable from N-Acetylcysteine, in addition to the medication regimen they are on at study enrollment.
  placebo : placebo, 2 capsules PO AM, 3 capsules PO PM, 6 weeks
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 4 | 2
Received Allocated Intervention | 3 | 2
Completed | 1 | 1
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Self-Harm Inventory (SHI) Score at 6 Weeks
Description: The Self-Harm Inventory is assessed by asking an individual to answer (yes or no) if they have ever "intentionally, or on purpose" tried to harm themselves. The inventory contains 22 questions and a 23rd marked "other" that allows the individual to indicate a self-harm behavior not previously mentioned.
  The scoring of this instrument is determined by counting the number of endorsed self-harm behaviors out of the possible twenty-three asked. The maximum score any individual may achieve for the SHI is a 23. Any individual scoring 5 or greater is classified as suffering from BPD.
  In this study, scoring on the SHI was primarily used to assess improvement of self-harming symptoms and throughout the study by comparing participant ratings from baseline and week 6. Positive numbers indicate a decrease (i.e. participant indicated less self-harming behavior) and negative numbers indicate an increase in self-harming behaviors reported.
Time Frame: 6 weeks
Measure: Number; unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | 5 | 1

2. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) at 6 Weeks
Description: The Hamilton Rating Scale for Depression is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. Administered by a clinician, The questionnaire is designed for adults and is used to rate the severity of the patients depression by asking their mood, feelings of guilt, insomnia, agitation, weight change, suicidal ideation, and somatic symptoms. The scale also allows the clinician to assess the patient's level of retardation, and insight into their depression. Highest possible score is 52.
  HAM-D Scoring 0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severed Depression
  ≥23 = Very Severe Depression
  In this study, Baseline ratings were compared to those of week 6 to assess each participants change in depression throughout the study. A negative value indicates an increase in depression (i.e. the individual felt more depressed) and a positive value indicates a decrease in depression.
Time Frame: 6 weeks
Measure: Number; unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | 28 | 18

3. Primary Outcome: Self-Harm Inventory (SHI) Score at Baseline
Description: as for outcome 1
Time Frame: Baseline
Measure: Number; unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | 8 | 4

4. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) at Baseline
Description: as for outcome 2
Time Frame: Baseline
Measure: Number; unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | 25 | 27

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes